CLINICAL TRIAL: NCT00129831
Title: Dose Escalation Study to Assess the Safety and Tolerability of Incremental Doses of QAB149 in Adults With Mild-to-moderate Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study to Assess the Safety and Tolerability of Incremental Doses of QAB149 in Adults With Mild-to-moderate Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQAB149B2202
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: COPD
Keywords: COPD, indacaterol, PK
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

INTERVENTIONS:
Drug: QAB149

SUMMARY:
The purpose of this study is to determine the safety and tolerability of single doses of QAB149 up to 3000 µg delivered via a single-dose, dry powder inhaler in patients with mild to moderate COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female patients with mild to moderate stable COPD, diagnosed according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines; 40-75 years of age
* Prebronchodilator baseline forced expiratory volume in 1 second (FEV1) 30-80% of the Quanjer predicted normal value (Quanjer et al. 1993) and at least 0.75 L with FEV1/forced vital capacity (FVC) < 70% of predicted [GOLD guidelines].
* Previous smokers (>10 pack-years). Ten pack years are defined as: 20 cigarettes a day for 10 years; 10 cigarettes a day for 20 years; or 40 cigarettes a day for 5 years. Current smokers, with >10 pack year history, can be included under certain conditions.
* Vital signs (after 3 minutes resting measured in the supine position) which are within the following ranges:

  * oral body temperature between 35.0-37.5 °C;
  * systolic blood pressure, 100-170 mm Hg;
  * diastolic blood pressure, 50-100 mm Hg;
  * pulse rate, 50 - 90 beats per minute (bpm).
* Patients must weigh a minimum of 50 kg to participate in this study.
* Able to provide written informed consent prior to study participation.
* Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion Criteria:

* Pregnant women or nursing mothers.
* Patients with a QTc interval above 0.43 seconds for males and 0.45 seconds for females at the screening visit. If pre-treatment values on Day 1 of the treatment periods exceed 0.45 and 0.47 seconds for males and females respectively the visit may be re-scheduled once.
* Patients with a history of prolonged QTc intervals, or a family history of prolonged QT syndrome.
* Predominant diagnosis of asthma. (Patients must present without evidence of active asthma.)
* Patients who have been hospitalized or had emergency treatment for acute COPD exacerbation in the one month prior to or during screening.
* Patients who have had a respiratory tract infection within one month prior to screening.
* Patients with concomitant pulmonary disease, including a history of cancer

Other exclusion criteria apply.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-09; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Safety variables (laboratory tests, ECG, adverse events)

SECONDARY OUTCOMES:
Lung function tests
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Radiant Research, Encinitas, California
  - Radiant Research, Boise, Idaho